CLINICAL TRIAL: NCT00223964
Title: Randomized Double-Blind Parallel Group MultiCenter Study of the Efficacy of Two Doses of Ferrlecit® in Treatment of Iron Deficiency in Pediatric Hemodialysis Patients Receiving Epoetin.
Brief Title: Study of the Efficacy of Two Doses of Ferrlecit in the Treatment of Iron Deficiency in Pediatric Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FR01006
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Anemia
Keywords: Iron Deficiency; Anemia in Pediatric Hemodialysis
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — ferric gluconate; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- dose level 1 (Experimental): 1.5 mg/kg
  Interventions: Drug: Ferrlecit (sodium ferric gluconate complex in sucrose injection)
- dose level 2 (Experimental): 3 mg/kg
  Interventions: Drug: Ferrlecit (sodium ferric gluconate complex in sucrose injection)

INTERVENTIONS:
Drug: Ferrlecit (sodium ferric gluconate complex in sucrose injection)

SUMMARY:
This was a multi-center study in iron-deficient pediatric hemodialysis patients, whose legal guardian had provided signed informed consent and satisfied the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric end-stage renal disease (ESRD) patients.
* Predetermined TSAT and serum ferritin levels
* Receiving chronic hemodialysis therapy with an identified need for repletion iron therapy.
* Receiving a stable epoetin (EPO) dosing regimen.

Exclusion Criteria:

* Receipt of any form of iron supplements during the 4 weeks prior to the first Ferrlecit® dosing.
* Blood transfusion.
* Hypersensitivity to Ferrlecit®.
* Significant inflammatory conditions.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2003-06; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Demonstrate and compare effectiveness of two Ferrlecit® doses in increasing hemoglobin in iron-deficient pediatric hemodialysis patients requiring repletion iron therapy. | 2 weeks

SECONDARY OUTCOMES:
Evaluate single-dose pharmacokinetics of Ferrlecit® in iron deficient pediatric hemodialysis patients and to access the safety profile of Ferrlecit® in pediatric hemodialysis patients. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GARY HOEL, RPh, PhD, Study Director — WATSON LPHARMACEUTICAL
Locations (24):
- United States (8):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Diego, California
  - Stanford, California
  - Boston, Massachusetts
  - Kansas City, Missouri
  - The Bronx, New York
  - Seattle, Washington
- Mexico (2):
  - Aruascalientes
  - Mexico City
- Poland (9):
  - Bialystok
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Szczecin
  - Torum
  - Wroclaw
  - Zabrze
- Russia (4):
  - Bashkortostan
  - Moscow
  - Saint Petersburg
  - Tartarstan
- Belgrade, Serbia